CLINICAL TRIAL: NCT04731662
Title: Effects of Recurrent Short and Variable Sleep on Cognitive Performance, Brain Dynamics, Psychological Well-being, and Glucose Metabolism
Brief Title: Performance, Mood, and Brain and Metabolic Functions During Different Sleep Schedules
Acronym: STAVAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Singapore (Other)
Responsible Party: Principal Investigator, June Chi Yan Lo, Principal Investigator, Assistant Professor, National University of Singapore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: STAVAR
Record Dates: First submitted 2021-01-26; First posted 2021-02-01 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Sleep; Sleep Restriction
Keywords: Glucose Metabolism; fMRI; Subjective Sleepiness; Neurobehavioral Functions; Cognitive Functions; Sleep Variability

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control Group (8888888) (No Intervention): The Control group will have 8-hours time-in-bed, both weeknights and weekends.
- Stable Short Sleep (8866666) (Experimental): The short sleep group will have 6-hours time-in-bed on weeknights and 8-hours time-in-bed on weekends.
  Interventions: Behavioral: Short sleep
- Variable short sleep group (8884846) (Experimental): The short sleep group time in-bed will vary across weeknights but will maintain the same amount of total time-in bed as the stable short sleep (8866666).
  Interventions: Behavioral: Variable short sleep

INTERVENTIONS:
Behavioral: Short sleep — 6-hours time-in-bed during weeknights
  Arms: Stable Short Sleep (8866666)
Behavioral: Variable short sleep — Variable hours of time-in bed during weeknights
  Arms: Variable short sleep group (8884846)

SUMMARY:
This proposed project will investigate whether a variable or a stable sleep schedule will be more effective in minimizing neurobehavioural and metabolic deficits when total sleep opportunity across two weeks is below the recommended sleep duration. In this laboratory-based, stay-in study, 60 young adults will be randomized into 1 of 3 groups. After 2 nights of 8-h time-in-bed (TIB) that simulate longer sleep opportunities typical of weekends, the stable short sleep group will have a 6-h TIB in each of the following 5 'weeknights' (8866666). The variable short sleep group (8884846) will also have a total TIB of 30h during the 'weeknights', although TIB varies across the 'weeknights'. The nightly TIB of the well-rested control group will be 8h (8888888). These manipulations will repeat in the second week, enabling the tracking of outcome measures during recurrent weeks of sleep restriction on 'weekdays' and extension on 'weekends'. A test battery assessing basic cognitive functions and mood will be administered 5 times a day. A long-term memory encoding task will be administered after week 1. A functional Magnetic Resonance Imaging (fMRI) brain scan, and an Oral Glucose Tolerance Test (OGTT) will be conducted after the second 'weekend' night and after the last 'weeknight' each week. Continuous glucose monitoring will be conducted throughout the experiment. Sleep will be measured every night with polysomnography.

DETAILED DESCRIPTION:
This proposed project will investigate whether a variable or a stable sleep schedule will be more effective in minimizing neurobehavioural and metabolic deficits when total sleep opportunity across two weeks is below the recommended sleep duration. This project involves young adults aged 21 - 35. For the two weeks leading up to the stay-in study, participants' sleep-wake patterns will be assessed via actigraphy and sleep diary. For the first week, participants will be asked to follow their habitual sleep schedule, while in the following week, the participants will be instructed to follow a specific sleep schedule with an 8-h sleep opportunity each night during the 7-night period with no napping allowed.

After the two weeks of actigraphy, participants will begin the 16-day in-lab protocol. Participants will be randomised into 1 of 3 groups. All the participants will have an 8-h sleep opportunity during the first two nights (baseline nights) that simulate longer sleep opportunities typical of weekends. During the next 5 'weeknights', the participant's sleep opportunities will be manipulated depending on their assigned group. The stable short sleep group will have a 6-h TIB in each of the following 5 'weeknights' (8866666). The variable short sleep group (8884846) will also have a total TIB of 30h during the 'weeknights', although TIB varies across the 'weeknights'. The nightly TIB of the well-rested control group will be 8h (8888888). The same sleep schedules will be implemented in the second week. The protocol will end with an 8-h sleep opportunity on night 15. For each participant, wake times will remain the same (i.e., participant's own habitual wake time derived from self-report and actigraphy) for all the TIBs. Thus, bedtimes will be delayed progressively with decreasing TIBs for the short sleep groups.

A battery of cognitive tests and psychological scales (approximately 30 minutes) will be administered 5 times a day at 3-hourly intervals, starting from 1.5 hours since awakening.

A memory encoding task will be administered on Day 8 to determine whether a variable/stable short sleep schedule is less disruptive to the acquisition of long-term memory. During the task, participants will be presented with 160 images containing a stimulus (e.g. landscapes) or no stimulus on a computer screen. Each image will be displayed for 2500ms followed by a response screen to prompt participants to indicate if a stimulus was previously presented. On Day 10, a randomized set of 240 images consisting of the 160 images previously shown (i.e. "old" images) and 80 "new" images will be presented to participants. Participants are tested on their recognition of the "old images" by selecting on a 5-point scale: (1) definitely did not see, (2) probably did not see), (3) unsure, (4) probably saw, (5) definitely saw. The two tasks will take approximately 25 minutes each.

An OGTT and fMRI brain scan will be performed after the second baseline night 2 (Day 3) and the last 'weeknight' each week (Day 8 and 15). Participants will be asked to perform 8 hours of overnight fasting before each OGTT. On the morning of the OGTT, an intravenous catheter will be inserted into the forearm of participants. Thereafter, 6 mL of blood samples will be drawn in a lying/sitting position. Participants will then be given a 75-g glucose solution to finish drinking within 7-10mins. 6 mL of blood samples will be collected again at time 15, 30, 60, and 120 minutes to measure for changes in glucose and insulin levels.

In addition to OGTT, the investigators will be using continuous glucose monitoring to measure glucose responses to the various sleep schedule throughout the 16-day study via a glucose sensor applied to the back of the participants' upper arms. To ensure the validity of the continuous glucose data, the investigators will provide three main meals each day to the participants, except on the OGTT days when only lunch and dinner will be provided. The portion of the food provided each day will ensure that each participant will consume the daily calorie and macronutrient requirement, and thus, the participant will not gain or lose weight during the study. Participants will be required to finish all the food provided.

During the fMRI brain scans, resting-state and task-related brain activity will be recorded. During part of the scan, participants will be required to perform the gradual onset continuous performance task (Esterman et al., 2013) wherein participants will be presented with grayscale photographs of different scenes (e.g. mountain and city scenes) in a random manner. Each scene is presented for 1600ms with a 800ms overlap with an interpolated transitions. Participants will then be instructed to press a button if a particular scene is identified (e.g. city scene), and withhold their responses to other scenes. Before the task, participants will be given the opportunity to get familiarised with the images and have a 1-minute practice session.

Sleep macro-structure (i.e., the duration of various sleep stages) and micro-structure (such as SWA) will be measured with polysomnography (PSG) every night. Electrodes will also be affixed to the participant's scalp for electroencephalographic (EEG) recording, around the eyes for electrooculographic (EOG) recording, under the chin for electromyographic (EMG) recording, and on the chest for electrocardiogram (ECG) recording. Pulse oximetry, a non-invasive method that employs a light sensor on a finger cuff, is used in the first baseline night for oxygen saturation measurement to verify that the participants do not suffer from sleep apnea.

Throughout the 16-day in-lab protocol, participants will not be allowed to leave the lab premises or engage in any strenuous exercise. When there are no research procedures being carried out, participants are free to spend their spare time on any activity, with the exception of napping, exercising, or activities that requires the participants to leave the lab premises. Participants will be under constant supervision by the research staff.

ELIGIBILITY:
Inclusion Criteria:

* 21-35 years of age
* Healthy
* BMI between 18.5 and 24.9
* Not habitual short sleepers
* Not extreme chronotypes
* Not a shift worker
* Not a smoker
* Daily consumption of ≤ 5 cups of caffeinated beverages
* Weekly consumption of ≤ 14 units of alcohol
* Do not intend to travel across > 2 time zones 1 month prior to the experiment
* Not a fussy eater
* Do not have any food allergy
* No strict dietary requirements
* No intention to lose or gain weight in the next 6 months
* Not pregnant during the study
* Do not have any metallic implants
* Do not suffer from claustrophobia (last three inclusion criteria are only applicable for fMRI)

Exclusion Criteria:

* The reverse of the inclusion criteria

Ages: 21 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-12-22 (Actual); Study Completion 2022-12-22 (Actual)

PRIMARY OUTCOMES:
Change in sustained attention assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 5 times daily for 16 days
  Number of attention lapses (>500ms)
Change in mean reaction time assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 5 times daily for 16 days
  Mean reaction time
Change in median reaction time assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 5 times daily for 16 days
  Median reaction time
Change in standard deviation in reaction time of sleep restriction and recovery | 5 times daily for 16 days
  Standard deviation in reaction time
Change in number of commission errors / false starts assessed with the Psychomotor Vigilance Task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep restriction and recovery | 5 times daily for 16 days
  Number of commission errors / false starts
Change in number of correct matches assessed with the 1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of correct matches in the 1-back task
Change in number of correct mismatches assessed with the1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of correct mismatches in the 1-back task
Change in number of incorrect matches assessed with the1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of incorrect matches in the 1-back task
Change in incorrect mismatches assessed with the1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of incorrect mismatches in the 1-back task
Change in discriminability measure (A') assessed with the1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Discriminability measure (A')
Change in bias measure (B"D) assessed with the1-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Bias measure (B"D)
Change in number of correct matches assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of correct matches in the 3-back task
Change in number of correct mismatches assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of correct mismatches in the 3-back task
Change in number of incorrect matches assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of incorrect matches in the 3-back task
Change in number of incorrect mismatches assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Number of incorrect mismatches in the 3-back task
Change in discriminability measure (A') assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Discriminability measure (A')
Change in bias measure (B"D) assessed with the 3-back task from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Bias measure (B"D)
Change in the level of subjective sleepiness assessed with the Karolinska Sleepiness Scale from morning to afternoon then evening from baseline days to the first and second cycle of sleep manipulation and recovery | 5 times daily for 16 days
  Score on the Karolinska Sleepiness Scale (1-9 points)
Change in positive mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Total score on the positive subscale of the PANAS
Change in negative mood assessed with the Positive and Negative Affect Scale (PANAS) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily for 16 days
  Total score on the negative subscale of the PANAS
Change in the level of depressive symptomatology from the mornings of the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 separate days (Day 3, 8 and 15)
  Score on the Mood and Anxiety Symptom Questionnaire (Scale 1-5)
Change in the level of anxiety symptomatology from the mornings of the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 separate days (Day 3, 8 and 15)
  Score on the Mood and Anxiety Symptom Questionnaire (Scale 1-5)
Change in the level of satisfaction with life from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily (09:00, 12:00, 15:00, 18:00, 21:00) for 16 days
  Score on the Satisfaction with Life Scale (1-7 scale)
Change in speed of processing assessed with the Mental Arithmetic Test (MAT) from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily (09:00, 12:00, 15:00, 18:00, 21:00) for 16 days
  Number of correct response in the task
Change in speed of processing assessed with the Symbol Digit Modalities Test from morning to afternoon and then evening from baseline days to the first and second cycles of sleep manipulation and recovery | 5 times daily (09:00, 12:00, 15:00, 18:00, 21:00) for 16 days
  Number of correct responses in the task
Changes in the blood glucose levels from morning of the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 days (Day 3, 8 and 15) 6mL blood sample collection at 15, 30, 60, and 120 minutes
  Area under the curve for plasma glucose
Changes in the insulin levels from morning of the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 days (Day 3, 8 and 15) 6mL blood sample collection at 15, 30, 60, and 120 minutes
  Area under the curve for insulin
Changes in interstitial fluid glucose levels from morning to afternoon then evening from baseline days to the first and second cycles of sleep manipulation and recovery. | All 16-days with 8-hour interval readings
  Area under the curve for interstitial fluid glucose
Changes in the task related brain functional connectivity from the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 days (Day 3, 8, 15)
  Brain functional connectivity in fMRI analysis
Changes in the resting-state brain functional connectivity from the second baseline day to the last day of the first sleep manipulation cycle and the last day of the second sleep manipulation cycle. | 3 days (Day 3, 8, 15)
  Brain functional connectivity in fMRI analysis
Effect of variable sleep on picture encoding response time | Single session (Day 8)
  Mean response time
Effect of variable sleep on picture encoding response accuracy | Single session (Day 8)
  Response accuracy
Effect of variable sleep on picture recognition response time | Single session (Day 10)
  Mean response time
Effect of variable sleep on picture recognition hit rate | Single session (Day 10)
  Hit rate
Effect of variable sleep on picture recognition false alarm rate | Single session (Day 10)
  False alarm rate
Effect of variable sleep on picture recognition discriminability measure (A') | Single session (Day 10)
  Discriminability measure (A')

SECONDARY OUTCOMES:
Change in total sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total duration of nocturnal sleep will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in wake after sleep onset duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total duration of wake after sleep onset will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change sleep efficiency at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total sleep efficiency will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change slow wave activity/ slow wave energy at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total slow wave activity/ slow wave energy will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change spindle activity at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total spindle activity will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in N1 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total duration of nocturnal N1 sleep duration will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in N1 sleep percentage at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Percentage of nocturnal N1 sleep duration will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in N2 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Duration of nocturnal N2 sleep will be determined to established baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)(first and second nights) and changes in the first sleep manipulation (third, forth, fifth, sixth
Change in N2 sleep percentage at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Percentage of nocturnal N2 sleep will be determined to established baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)(first and second nights) and changes in the first sleep manipulation (third, forth, fifth, sixth
Change in N2 sleep latency at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Duration of nocturnal N2 sleep latency will be determined to established baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)(first and second nights) and changes in the first sleep manipulation (third, forth, fifth, sixth
Change in N3 sleep duration at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Total duration of nocturnal N3 sleep will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth, and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in N3 sleep percentage at night assessed with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Percentage of nocturnal N3 sleep will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth, and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in the Rapid Eye Movement (REM) sleep duration at night with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Duration of nocturnal sleep REM sleep will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)
Change in the Rapid Eye Movement (REM) sleep percentage at night with polysomnography from baseline nights to the first and second cycles of sleep manipulation and recovery | Nocturnal sleep on nights 1 & 2 (baseline), 3, 4, 5, 6 & 7 (first sleep manipulation period), 8 & 9 (first recovery period), 10,11,12, 13, 14 (second sleep manipulation period), & 15 (second recovery period)
  Percentage of nocturnal sleep REM sleep will be determined to establish baseline sleep characteristics (first and second night) and changes in the first sleep manipulation period (third, fourth, fifth, sixth and seventh sleep) the first recovery period (eight and ninth night), the second sleep manipulation period (tenth, eleventh, twelfth, thirteenth, fourteenth), and the second recovery period (15th night)

CONTACTS AND LOCATIONS:
Overall Officials: June Chi Yan Lo, Principal Investigator — National University of Singapore
Locations (1):
- MD 11- NUS Yong Loo Lin School of Medicine, Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cheung YYY, Tan TYL, Koa TB, Khoo CM, Lo JC. Glucose homeostasis during recurrent periods of sleep restriction and recovery in healthy young adults. Sleep. 2025 Oct 30:zsaf339. doi: 10.1093/sleep/zsaf339. Online ahead of print. PMID 41165770
- [Derived] Koa TB, Ong JL, Lo JC. Changes in sleep architecture during recurrent cycles of sleep restriction: a comparison between stable and variable short sleep schedules. Sleep Adv. 2025 Mar 15;6(2):zpaf016. doi: 10.1093/sleepadvances/zpaf016. eCollection 2025 Apr. PMID 40385325
- [Derived] Koa TB, Gooley JJ, Chee MWL, Lo JC. Neurobehavioral functions during recurrent periods of sleep restriction: effects of intra-individual variability in sleep duration. Sleep. 2024 Mar 11;47(3):zsae010. doi: 10.1093/sleep/zsae010. PMID 38219041